CLINICAL TRIAL: NCT02969278
Title: Study on the Prediction of Groin Lymphonodal Status Through 18FDG-PET/CT Combined With Sentinel Lymph Node Biopsy in Bulky a/o Multifocal a/o Pretreated Vulvar Cancer, N0 at Conventional Imaging (GRO-SNaPET Study)
Brief Title: Groin Sentinel Node Biopsy and 18FDG-PET/CT in cN0 Vulvar Cancer Patients Candidate to Standard Lymphadenectomy
Acronym: GroSNaPET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GroSNaPET
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Vulvar Cancer
Keywords: vulvar cancer; sentinel node biopsy; inguino-femoral lymphadenectomy; 18F FDG- PET/TC; guidelines; preoperative imaging
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vulvar cancer patients cN0 unfit for sentinel node biopsy (Experimental): All invasive vulvar cancer patients with cN0 status:
  * T > 4 cm;
  * multicentric tumors (mono or bilateral);
  * primary lesion completely excised during prior diagnostic surgery
  * patients candidate to bilateral lymphadenectomy because of unilateral groin lymph node involvement, contralateral cN0
  * previous radiotherapy a/o chemotherapy (sequential or concurrent). These patients are submitted to 18FDG PET/TC and sentinel node biopsy associated with standard preoperative imaging and radical groin lymphadenectomy
  Interventions: Procedure: 18FDG-PET/TC; Procedure: Sentinel node biopsy

INTERVENTIONS:
Procedure: 18FDG-PET/TC — Nuclear medicine exam (18FDG-PET/TC) to assess the status of the regional groin and pelvic lymphnodes
Procedure: Sentinel node biopsy — Intradermal injection of 0.2 ml 37-148 MBq of radiocolloid and a blue dye near the tumor to locate the position of the sentinel lymph node. Intraoperatively, sentinel node localization is guided by a gamma probe and by the eyes of the surgeon who detects the lymph nodes that are stained with the blue dye.

SUMMARY:
The study aim is to verify the accuracy of SNB combined with 18F-FDG PET/CT in cN0 invasive vulvar cancer (IVC) patients currently not candidate to SNB according to standard guidelines.

DETAILED DESCRIPTION:
Vulvar carcinoma (VC) is a rare disease (4% of gynecological cancers) and the treatment is not yet universally defined. No official guidelines are currently available to define imaging techniques useful for staging. In the pre-operative evaluation of the pateints, imaging should assess nodal status; the available exams are:

* CT or MRI with contrast (abdominal and pelvic with caudal scans for inguinal regions)
* Inguinal ultrasound with US-guided biopsy/fine needle aspiration for suspicious lymph nodes.

The incidence of inguinal and pelvic lymph node metastasis not diagnosed at the pre-operative imaging is 10-35% as assessed after lymphadenectomy at pathology report.

Until 2009, the standard surgical treatment of vulvar cancer was represented by mono or bilateral systematic lymphadenectomy (at least 70% of N0 women underwent a radical surgery with the risk of severe morbidity related to the surgical procedure with no survival benefit).

Inguinal lymphadenectomy shows a high rate of local and systemic complications resulting in a longer hospitalization or recovery, as well as possible delays in adjuvant therapies.

Moreover, severe complications can lead to a further surgery.

Possibile complications described in literature are:

* Lymphedema (up to 70%)
* Infection and postoperative cellulitis (50%)
* Inguinal suture dehiscence (between 22 and 52%)
* Linfocysts (between 7 and 28%)
* Deep vein thrombosis (between 5 and 8%)
* Sepsis (1 -2%)

Since 2009, with the introduction and the validation of sentinel node biopsy (SNB), for some VC it is now possible to obtain a nodal staging with minimally invasive surgery and lower morbidity. However, the SNB technique is indicated if the tumor fits the following selection criteria:

* Infiltrating tumors with a diameter < 40 mm;
* Monofocal tumors;
* Tumors distant more than 1 cm from the midline
* Tumors near the midline with bilateral lymphatic drainage and intraoperative detection of at least one sentinel node for each groin.

Consequently in many tumors diagnosed as N0 at preoperative imaging, SNB technique is not indicated; these tumors still require systematic lymphadenectomy.

In this subset of patients it is important to identify new methods for preoperative evaluation of nodal status or to define a sub-category of patients for which the SNB could be applied.

Objective of the study is to verify, in patients actually off-label for SNB, the accuracy of 18FDG-PET/CT in predicting nodal status, as an indipendent method or associated with the standard pre-operative imaging and the mini-invasive surgical staging.

All patients are submitted to:

* Gynecologic visit
* Vulvar biopsy and possible pelvic examination under anesthesia with the definition of clinical extent of disease
* Evaluation of serum tumor markers: SCC and Ca125
* Inguinal ultrasound and possible US guided FNAC or FNAB on suspicious lymph nodes
* CT scan (abdomen and pelvis) with contrast
* 18FDG-PET/CT
* Lymphangioscintigraphy of inguinofemoral axis

Vulvar surgery may include:

* Wide resection of vulvar disease
* Emivulvectomy (anterior, posterior or lateral)
* Simple vulvectomy
* Radical or ultra-radical vulvectomy (with possible plastic reconstruction)

During inguinal surgery all patients will undergo:

- Sentinel node biopsy mono or bilateral followed by radical bilateral inguinal lymphadenectomy

Statistical analysis will help determine the accuracy and negative predictive value of FDG-PET/CT and sentinel node biopsy in predicting nodal status.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* ECOG ≤ 2
* Adequate respiratory, hepatic, cardiac, bone marrow and renal function (creatinine clearance> 60 mL/min according to the Cockroft formula)
* Patient psychologically able to follow the study procedures
* Signature of informed consent

In addition, both major criteria and at least one of the minor criteria must be present:

MAJOR CRITERIA

* Vulvar carcinoma (stromal infiltration > 1 mm); Histotypes different from squamous are included
* Negative lymphnodes at preoperative imaging

MINOR CRITERIA

* Vulvar lesion greater than 4 cm
* Multifocal or bilateral lesions
* Previous complete excisional biopsy of the vulvar lesion, with absent residual disease
* Previous neoadjuvant treatment (radiotherapy a/o sequential/concomitant chemotherapy)
* Previous treatment with radiotherapy a/o chemotherapy (sequential a/o concomitant) for previous vulvar cancer a/o other diseases
* Previous vulvar or inguinal surgery
* Infiltrating vulvar carcinoma with monolateral groin lymphnode involvement (N1) and contralateral N0

Exclusion Criteria:

* Allergy to egg proteins and albumin
* Pregnancy and breastfeeding
* Patients with impaired respiratory, hepatic, cardiac, bone marrow and renal function (creatinine clearance> 60 mL / min according to the Cockroft formula)
* Patients with major depressive disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy and Negative Predictive Value of sentinel node biopsy in cN0 vulvar cancer patients that do not fit for the current indications | within the first 30 days after surgery

SECONDARY OUTCOMES:
Accuracy and Negative Predictive Value of preoperative 18F FDG-PET/CT for the selection of cN0 patients. | within the first 60 days before surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gynecologic Oncology/Fondazione Policlinico Gemelli, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No